CLINICAL TRIAL: NCT04747808
Title: A Phase 2a Study of Safety, Tolerability, and Efficacy of Drug-Delivering Contact Lens LL-BMT1 in Patients With Primary Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Study of LL-BMT1 in Patients With Elevated Intraocular Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MediPrint Ophthalmics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LL-BMT10001
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Results first posted 2022-05-10 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-04

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Prostaglandin; Intraocular pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma

STUDY DESIGN:
Intervention Model Description: Open-label, non-comparative
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LL-BMT1 (Experimental): Group 4 extended-wear contact lens printed with bimatoprost
  Interventions: Drug: LL-BMT1

INTERVENTIONS:
Drug: LL-BMT1 — Drug-printed contact lens in both eyes

SUMMARY:
This is an open-label, Phase 2a clinical study of LL-BMT1 in patients with primary open-angle glaucoma and ocular hypertension. Study subjects will be treated for 7 days with a single dose of LL-BMT1.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age at the Screening Visit
* Diagnosed with primary open-angle glaucoma or ocular hypertension in both eyes
* At least one eye (called the study eye) must have an untreated intraocular pressure between 22 mmHg and 34 mmHg (inclusive) as measured at 9 am during the Baseline Visit.
* Best corrected visual acuity of Early Treatment Diabetic Retinopathy Study of 50 letters or better

Exclusion Criteria:

* Glaucoma or optic neuropathy due to anything other than above noted reasons Cup-to-disc ratio of >0.8 in either eye
* Corneal thickness <480 or >620 μm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Research Foundatoin, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LL-BMT1
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LL-BMT1
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.4 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Intraocular pressure (study eye) [Mean (Standard Deviation); unit: mm Hg] | 24.7 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Adverse Event Rate
Description: Number of subjects with adverse events
Time Frame: Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | LL-BMT1
Number analyzed (Participants) | 5
Participants | 1

2. Secondary Outcome: Intraocular Pressure Elevation
Description: Number of subjects with IOP elevation >= 5 mm Hg in study eye
Time Frame: Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | LL-BMT1
Number analyzed (Participants) | 5
Participants | 0

3. Secondary Outcome: IOP Changes
Description: Mean change in IOP from baseline in study eye (mm Hg) on Day 1, 4 pm
Time Frame: Days 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LL-BMT1
Number analyzed (Participants) | 5
mmHg | -2.9 (0.7)

ADVERSE EVENTS:
Time Frame: 8 Days
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | LL-BMT1
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 1/5
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LL-BMT1 (N=5)
Ocular irritation (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT04747808/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/08/NCT04747808/SAP_001.pdf